CLINICAL TRIAL: NCT06297616
Title: A Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3841136 Monotherapy, and LY3841136 in Combination With Tirzepatide, in Japanese Participants With Obesity or Overweight
Brief Title: A Study of LY3841136 in Japanese Participants With Obesity or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18814; J3R-JE-YDAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
Keywords: Obesity Disease; Metabolic Disorders; Body Weight Loss
MeSH Terms: conditions — Obesity; Overweight; Metabolic Diseases | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part A: LY3841136 (Experimental): LY3841136 administered subcutaneously (SC)
  Interventions: Drug: LY3841136
- Part A: Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: LY3841136-Placebo
- Part B: Tirzepatide + LY3841136-Placebo (Experimental): Tirzepatide administered SC along with volume-matched LY3841136-Placebo administered SC
  Interventions: Drug: LY3841136-Placebo; Drug: Tirzepatide
- Part B: LY3841136 + Tirzepatide-Placebo (Experimental): LY3841136 administered SC along with volume-matched Tirzepatide-Placebo administered SC
  Interventions: Drug: LY3841136; Drug: Tirzepatide-Placebo
- Part B: LY3841136 + Tirzepatide (Experimental): LY3841136 administered SC along with Tirzepatide administered SC
  Interventions: Drug: LY3841136; Drug: Tirzepatide
- Part B: LY3841136-Placebo + Tirzepatide-Placebo (Placebo Comparator): Volume-matched LY3841136-Placebo administered SC along with volume-matched Tirzepatide-Placebo administered SC
  Interventions: Drug: LY3841136-Placebo; Drug: Tirzepatide-Placebo

INTERVENTIONS:
Drug: LY3841136 — Administered SC
  Arms: Part A: LY3841136; Part B: LY3841136 + Tirzepatide; Part B: LY3841136 + Tirzepatide-Placebo
Drug: LY3841136-Placebo — Administered SC
  Arms: Part A: Placebo; Part B: LY3841136-Placebo + Tirzepatide-Placebo; Part B: Tirzepatide + LY3841136-Placebo
Drug: Tirzepatide — Administered SC
  Arms: Part B: LY3841136 + Tirzepatide; Part B: Tirzepatide + LY3841136-Placebo
Drug: Tirzepatide-Placebo — Administered SC
  Arms: Part B: LY3841136 + Tirzepatide-Placebo; Part B: LY3841136-Placebo + Tirzepatide-Placebo

SUMMARY:
The main purpose of this study is to learn about the side effects of LY3841136 alone and in combination with tirzepatide, when given to Japanese participants with obese or overweight. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. Part A of the study will last about 28 weeks and may include up to 17 visits. Part B of the study will last about 40 weeks and may include up to 29 visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who agree to contraception requirements
* Have a body mass index (BMI) within the range of 27 to 40 kg/m², inclusive
* Have had a stable weight for the 3 months

Exclusion Criteria:

* Have a history of significant atopy (severe allergic manifestations), multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions
* Have a history or presence of psychiatric disorders, including a history of major depressive disorder or severe psychiatric disorders such as schizophrenia, bipolar disorder within the last 3 years
* Have been diagnosed with Type 1 or Type 2 Diabetes Mellitus
* Have a history of chronic medical conditions involving the heart, liver, or kidneys
* Have a history of any malignancy within the past 5 years
* Have a history or presence of a GI disorder
* Have had within the last 6 months, or plan to have during the study, a device-based or surgical treatment use for obesity
* Have been treated, or plan to be treated, with prescription medications or other non-approved drugs intended to promote weight loss, within 3 months prior to screening
* For participants in Part B, have previously received tirzepatide within 6 months prior to screening
* For participants in Part B, have a personal or family history of medullary thyroid carcinoma, or have multiple endocrine neoplasia syndrome type 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with One or More Serious Adverse Events (SAE) Considered by the Investigator to be Related to Study Drug Administration at Week 22 | Baseline through Week 22
  A summary of treatment emergent adverse events (TEAEs), SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Part B: Number of Participants with One or More Serious Adverse Events (SAE) Considered by the Investigator to be Related to Study Drug Administration at Week 34 | Baseline through Week 34
  A summary of treatment emergent adverse events (TEAEs), SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Part A Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3841136 | Predose through Week 22
  PK: AUC of LY3841136 alone
Part A PK: Maximum Observed Concentration (Cmax) of LY3841136 | Predose through Week 22
  PK: Cmax of LY3841136 alone
Part A Pharmacodynamics (PD): Change From Baseline in Body Weight at Week 12 | Baseline through Week 12
  PD: Change from baseline in body weight
Part B PK: AUC of LY3841136 in Combination with Tirzepatide | Predose through Week 34
  PK: AUC of LY3841136 in combination with tirzepatide
Part B PK: Cmax of LY3841136 in Combination with Tirzepatide | Predose through Week 34
  PK: Cmax of LY3841136 in combination with tirzepatide
Part B PD: Change From Baseline in Body Weight at Week 24 | Baseline through Week 24
  PD: Change from baseline in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (3):
  - P-One Clinic, Hachiōji, Tokyo
  - Sumida Hospital, Sumida-ku, Tokyo
  - Hakata Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3841136 in Japanese Participants with Obesity or Overweight — https://trials.lilly.com/en-US/trial/466940